CLINICAL TRIAL: NCT02912702
Title: A Randomized Controlled Trial of L-DEP as an Initial Treatment for Epstein-Barr Virus-associated Hemophagocytic Lymphohistiocytosis
Brief Title: L-DEP as an Initial Treatment for EBV-HLH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Doctor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-DEP-EBV-HLH-First line
Record Dates: First submitted 2016-09-09; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Pegaspargase; hemophagocytic lymphohistiocytosis; Epstein Barr virus; initial treatment
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections | interventions — pegaspargase; Etoposide; Methylprednisolone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-DEP (Experimental): Pegaspargase 2000U/m2 day5; doxorubicin hydrochloride liposome injection 25 mg/m2 day 1; etoposide 100 mg/m2 was administered once on the first day of every week; methylprednisolone 15 mg/kg days 1 to 3, 0.75 mg/kg days 4 to 7
  Interventions: Drug: Pegaspargase; Drug: doxorubicin hydrochloride liposome injection; Drug: etoposide; Drug: methylprednisolone
- HLH-94 regimen (Active Comparator): Etoposide 150 mg/m2 twice weekly for 2 weeks and then weekly; dexamethasone initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering
  Interventions: Drug: Etoposide; Drug: dexamethasone

INTERVENTIONS:
Drug: Pegaspargase — 2000U/m2 day5
  Arms: L-DEP
Drug: doxorubicin hydrochloride liposome injection — 25 mg/m2 day 1
  Arms: L-DEP
Drug: etoposide — 100 mg/m2 was administered once on the first day of every week
  Arms: L-DEP
Drug: methylprednisolone — 15 mg/kg days 1 to 3, 0.75 mg/kg days 4 to 7
  Arms: L-DEP
Drug: Etoposide — 150 mg/m2 twice weekly for 2 weeks and then weekly
  Arms: HLH-94 regimen
Drug: dexamethasone — initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering
  Arms: HLH-94 regimen

SUMMARY:
This study aimed to investigate the efficacy and safety of Pegaspargase together with liposomal doxorubicin, etoposide and high dose methylprednisolone (L-DEP) as an initial treatment for Epstein Barr virus-induced hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were older than 14 years of age
2. Diagnosed as EBV-Hemophagocytic Lymphohistiocytosis (HLH)
3. Patients did not receive any treatment for HLH before
4. Informed consent

Exclusion Criteria:

1. Heart function above grade II (NYHA)
2. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2
3. Pregnancy or lactating Women
4. Allergic to Pegaspargase, doxorubicin or etoposide
5. Active bleeding of the internal organs
6. uncontrollable infection
7. history of acute and chronic pancreatitis
8. Participate in other clinical research at the same time

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Overall response(complete response+ partial response) rate of Participants | Change from before and 2,4,6 and 8 weeks after initiating L-DEP or HLH-94 therapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25(pg/ml), ferritin(μg/L), and triglyceride(mmol/L); hemoglobin(g/L); neutrophil counts(×109/L); platelet counts(×109/L); and alanine aminotransferase (ALT(U/L)).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25(pg/ml) response was>1.5-fold decreased; ferritin (μg/L)and triglyceride(mmol/L) decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT (U/L)decrease of at least 50%.

SECONDARY OUTCOMES:
Compare survival between two arms | from the time patients received L-DEP or HLH-94 therapy up to 12 months or September 2019
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 years
  Adverse events including pancreatitis, liver function damage, myelosuppression, infection, bleeding and so on.
Change of Epstein-Barr virus(EBV)-DNA before and after therapy | Change from before and 2, 4, 6 and 8 weeks after initiating L-DEP or HLH-94 therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Y, Huang W, Hu L, Cen X, Li L, Wang J, Shen J, Wei N, Wang Z. Multicenter study of combination DEP regimen as a salvage therapy for adult refractory hemophagocytic lymphohistiocytosis. Blood. 2015 Nov 5;126(19):2186-92. doi: 10.1182/blood-2015-05-644914. Epub 2015 Aug 19. PMID 26289641